CLINICAL TRIAL: NCT03736499
Title: Endocrine Changes in Adults Undergoing Cardiac Surgery
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Semmelweis University Heart and Vascular Center (Other)
Responsible Party: Principal Investigator, Andrea Szekely, Associate Professor, Semmelweis University Heart and Vascular Center
Other Study IDs: SE VSZÉK EndocrinHeart
Record Dates: First submitted 2018-10-25; First posted 2018-11-09 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2022-01

CONDITIONS: Endocrine System Diseases; Cardiac Surgery; Quality of Life; Psychology, Social
MeSH Terms: conditions — Endocrine System Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In this prospective study the investigators want to measure the serum level changes of the thyroid hormones (thyroid-stimulating hormone, reverse triiodothyronine, serum free T4), brain natriuretic peptide (BNP), testosterone and sexual hormone binding protein (SHBG) in adults undergoing cardiac surgery and search for correlations different psychosocial factors and analyze the influence on the survival and the length of ICU/hospital stay.

DETAILED DESCRIPTION:
In this study the investigators want to analyze routinely collected data of patients who underwent any kind of elective cardiac surgery in our university cardiovascular centre between 07.01.2018 and 30.06.2020. The database contains descriptive parameters, history of past illnesses, recent medication. The investigators record the type of surgery, the list of contributory physicians, the length of the surgery and the data of the anaesthesiological report. After the surgery the researchers want to record the postoperative parameters on the ICU ( infusion - fluid balance, blood transfusion, bleeding, main hemodynamic parameters, length of mechanical ventilation,main parameters of arterial blood gas analysis). Moreover th investigators want to collect psychosocial tests (Beck Depression Inventory, State Anxiety Scale, Trait Anxiety Scale and EQ-5D for the measurement of quality of life) to get more information from the postoperative condition of the patients.

ELIGIBILITY:
Inclusion Criteria:

* elective cardiac surgery

Exclusion Criteria:

* lack of consent
* pregnancy
* acute surgery
* exposition with iodin-containing contrast material

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 500 patients of a regional cardiovascular surgery centre
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2018-07-01 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2022-05-30 (Estimated)

PRIMARY OUTCOMES:
Length of hospital and intensive care unit stay | Participants will be followed for the duration of hospital stay, an expected average of 2 weeks.
  The correlation of the measured pre and postoperative endocrine profile and the length of intensive care unit stay

SECONDARY OUTCOMES:
The composite of in-hospital death from any cause. | Participants will be followed for the duration of hospital stay, an expected average of 12 weeks.
  Any cause of death in current group
Correlation between preoperative Beck Depression Inventory and the length of hospital stay | Participants will be followed for the duration of hospital stay, an expected average of 12 weeks.
  The effect of psychological state of the length of hospital stay
Correlation between preoperative State Anxiety Scale and the length of hospital stay | Participants will be followed for the duration of hospital stay, an expected average of 12 weeks.
  The effect of psychological state of the length of hospital stay
Correlation between preoperative Trait Anxiety Scale and the length of hospital stay | Participants will be followed for the duration of hospital stay, an expected average of 12 weeks.
  The effect of psychological state of the length of hospital stay
Correlation between preoperative EQ-5D inventory and the length of total hospital stay | Participants will be followed for the duration of hospital stay, an expected average of 12 weeks.
  Correlation between the preoperative quality of life state and the hospital stay

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Székely, ass. prof, Study Director — Semmelweis Egyetem; Ágnes Sándor, PhD st, Principal Investigator — Semmelweis Egyetem; András Szabó, PhD st, Principal Investigator — Semmelweis Egyetem
Locations (3):
- Hungary (3):
  - Heart and Vascular Center, Semmelweis University, Budapest
  - Semmelweis Egyetem Heart and Vascular Center, Budapest
  - Semmeweis Egyetem Heart and Vascular Center, Budapest

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Aversa A, Fabbri A. Testicular and thyroid function as survival predictors in the elderly patient candidate to surgery. Monaldi Arch Chest Dis. 2017 Jul 18;87(2):841. doi: 10.4081/monaldi.2017.841. PMID 28967725
- [Background] Brozaitiene J, Mickuviene N, Podlipskyte A, Burkauskas J, Bunevicius R. Relationship and prognostic importance of thyroid hormone and N-terminal pro-B-Type natriuretic peptide for patients after acute coronary syndromes: a longitudinal observational study. BMC Cardiovasc Disord. 2016 Feb 18;16:45. doi: 10.1186/s12872-016-0226-2. PMID 26892923
- [Background] Bianchi V, Mezzani A. Androgens and cardiac diseases. Monaldi Arch Chest Dis. 2013 Dec;80(4):161-9. doi: 10.4081/monaldi.2013.5232. PMID 25087292
- [Background] Maggio M, Nicolini F, Cattabiani C, Beghi C, Gherli T, Schwartz RS, Valenti G, Ceda GP. Effects of testosterone supplementation on clinical and rehabilitative outcomes in older men undergoing on-pump CABG. Contemp Clin Trials. 2012 Jul;33(4):730-8. doi: 10.1016/j.cct.2012.02.019. Epub 2012 Mar 5. PMID 22414875
- [Background] Fleischer J, McMahon DJ, Hembree W, Addesso V, Longcope C, Shane E. Serum testosterone levels after cardiac transplantation. Transplantation. 2008 Mar 27;85(6):834-9. doi: 10.1097/TP.0b013e318166ac10. PMID 18360264
- [Background] Kunst G, Pfeilschifter J, Kummermehr G, Luntz S, Bauer H, Martin E, Motsch J. Assessment of sex hormone-binding globulin and osteocalcin in patients undergoing coronary artery bypass graft surgery. J Cardiothorac Vasc Anesth. 2000 Oct;14(5):546-52. doi: 10.1053/jcan.2000.9450. PMID 11052436
- [Result] Razvi S, Jabbar A, Pingitore A, Danzi S, Biondi B, Klein I, Peeters R, Zaman A, Iervasi G. Thyroid Hormones and Cardiovascular Function and Diseases. J Am Coll Cardiol. 2018 Apr 24;71(16):1781-1796. doi: 10.1016/j.jacc.2018.02.045. PMID 29673469
- [Derived] Szecsi B, Toth K, Szabo A, Eke C, Szentgroti R, Dohan O, Benke K, Radovits T, Polos M, Merkely B, Gal J, Szekely A. Hormonal changes in the first 24 postoperative hours after cardiac surgical procedures. Physiol Int. 2023 Aug 4;110(3):251-266. doi: 10.1556/2060.2023.00219. Print 2023 Sep 5. PMID 37540593
- [Derived] Toth K, Szabo A, Menyhard J, Benke K, Radovits T, Polos M, Merkely B, Gal J, Szekely A. Poor Preoperative Nutritional Status, but Not Hormone Levels, Are Associated With Mortality After Cardiac Surgery. J Cardiothorac Vasc Anesth. 2022 Aug;36(8 Pt B):3074-3083. doi: 10.1053/j.jvca.2022.04.035. Epub 2022 Apr 29. PMID 35610144